CLINICAL TRIAL: NCT02733393
Title: Sphenopalatine Ganglion Block to Treat Shoulder Pain After Thoracotomy- An Open Label Pilot Study
Brief Title: Sphenopalatine Ganglion Block to Treat Shoulder Pain After Thoracotomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00618
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Ipsilateral Shoulder Pain
Keywords: Thoracotomy; Postoperative; Lidocaine; Sphenopalatine Ganglion Block
MeSH Terms: interventions — spirogermanium; Dental Occlusion; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SPG Block (Experimental)
  Interventions: Procedure: Sphenopalatine Ganglion (SPG) Block; Drug: lidocaine

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion (SPG) Block — Patients who are undergoing a thoracotomy will be informed that they may develop moderate to severe postoperative ISP and may have the option to receive an SPG block. The SPG block will be performed every three minutes for 20 minutes, 0.1mL of the 4% lidocaine will be administered through. After 20 minutes and various intervals thereafter the patient will be asked to rate their shoulder pain.
Drug: lidocaine

SUMMARY:
The purpose of this pilot study is to evaluate the utility of sphenopalatine ganglion (SPG) block to manage ipsilateral shoulder pain (ISP) after thoracotomy. This will be an open label preliminary pilot study to determine if SPG block has potential utility to manage ISP in post-thoracotomy patients. The primary outcome variable will be reduction of shoulder pain.

DETAILED DESCRIPTION:
This is an open label preliminary pilot study which will evaluate the utility of sphenopalatine ganglion (SPG) block to manage ipsilateral shoulder pain (ISP). It will determine if SPG block has potential utility to manage ISP in post-thoracotomy patients One hundred (100) patients will initially be consented in this study. Patients have to develop ISP and have a pain VAS >= 5. The study is seeking ten (10) eligible participants.

Patients will be followed after the SPG block(s), and the duration of pain relief will be monitored by serial assessments of the VAS. This assessment will occur for the initial SPG block and for all follow-up blocks, if performed. The follow-up assessments will only involve having the patient rate the ISP using a verbal VAS; This will take less than a minute of patients time. In addition, all patients will have PRN access to standard systemic analgesics as routinely ordered by the surgical service Safety assessments will be performed on all subjects. Blood pressure, heart rate and respiratory rate will be obtained every 15 minutes after each SPG block for 90 minutes. Dr. Grant will monitor the subjects for 90 minutes after each SPG block.

ELIGIBILITY:
Inclusion Criteria:

* Any type of open thoracotomy or video-assisted thoracoscopic surgery (VATS)
* Presence of post-operative ISP, VAS>5/10
* American Society of Anesthesiologists Class 1 - 4
* No allergy to lidocaine

Exclusion Criteria:

* American Society of Anesthesiologists Class 5
* Allergy to lidocaine
* Nasal pathology (e.g., deviated septum)
* Bleeding diathesis
* Any patient who the PI feels will be unable to comply with all protocol related procedures
* Shoulder pain prior to thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain Reduction | 90 Minutes
  Patients will be followed after the SPG block(s) and the duration of pain relief will be monitored by serial assessments of the VAS. This assessment will occur for the initial SPG block and for all follow-up blocks, if performed.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Grant, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States